CLINICAL TRIAL: NCT07406828
Title: Single Dose Psilocybin for a Post-surgical Trauma Inpatient Population for Pain, Mood, and Opioid Use Disorder
Brief Title: Psilocybin After Trauma Surgery for Pain
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Trent Emerick (Other)
Collaborators: The Beckwith Institute (Other)
Responsible Party: Sponsor-Investigator, Trent Emerick, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY24040071
Record Dates: First submitted 2026-01-31; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Pain Management; Postoperative Pain
Keywords: psilocybin; postoperative trauma; opioid; opioid use prevention; surgery; mushrooms; opioid adverse events
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Postoperative Standard of Care (Active Comparator): Participants receive standard postoperative pain management following trauma surgery, including multimodal analgesia and medications for opioid use disorder, as determined by the clinical care team. No psilocybin is administered.
  Interventions: Drug: Postoperative analgesia
- Single Dose Psilocybin (Experimental): Participants receive a single oral dose of psilocybin (10 mg) administered during inpatient hospitalization within 72 hours after trauma surgery, along with the standard postoperative care.
  Interventions: Drug: Psilocybin (Usona Institute); Drug: Postoperative analgesia

INTERVENTIONS:
Drug: Psilocybin (Usona Institute) — Single oral dose of psilocybin (10 mg) administered once during inpatient hospitalization to postoperative trauma surgery patients with opioid use disorder, followed by an 8-hour monitored observation period.
  Arms: Single Dose Psilocybin
Drug: Postoperative analgesia — Standard postoperative pain management, including multimodal analgesia and medications for opioid use disorder, provided per institutional clinical practice.

SUMMARY:
The goal of this clinical trial is to evaluate whether a single dose of psilocybin is feasible and safe for adults with opioid use disorder (OUD) who are recovering from trauma surgery. The main questions it aims to answer are:

1. Is a single psilocybin dose feasible to administer during postoperative hospitalization?
2. Is psilocybin safe in this patient population?
3. How does psilocybin affect postoperative pain, opioid use, anxiety, and depression after hospital discharge?

Participants will:

Receive one oral dose of psilocybin during their postoperative inpatient stay Complete assessments of pain, mood, and opioid use during recovery

DETAILED DESCRIPTION:
This is an open-label pilot feasibility trial conducted at a single academic medical center. Fourteen participants receive a single oral dose of psilocybin during inpatient hospitalization following trauma surgery. Outcomes in the psilocybin group are compared with a retrospectively identified standard-of-care cohort of 56 trauma surgery patients with opioid use disorder, identified through electronic medical record review.

The standard-of-care cohort is selected using propensity score methods based on baseline characteristics, including age, sex, trauma diagnosis, psychiatric comorbidities, baseline medications, comorbid conditions, type of surgery, and baseline opioid consumption measured in morphine milligram equivalents.

No interim efficacy analyses are planned. After the first three participants have received psilocybin and completed the one-week follow-up assessments, the Data and Safety Monitoring Board reviews safety data to assess ongoing risk and determine whether study procedures should continue unchanged.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 25 years old and ≤65 years old
2. Inpatient
3. English-speaking
4. History of opioid use disorder as diagnosed by DSM-V
5. Able to swallow capsules.
6. Patients are able to be enrolled and receive psilocybin within 3 days (72 hours) of surgery (time point 0 for this three-day window begins after patient arrival in the ICU) after a trauma surgery. Psilocybin will be administered in the morning to allow for the 8-hour monitoring period.

Exclusion Criteria:

1. Pregnancy. Women of child-bearing potential need to have a negative pregnancy test result at screening and baseline.
2. Sexually active male participants and/or their female partners and female participants of child-bearing potential need to be on adequate and effective method of contraception (diaphragm, male condom, combined pill, copper IUD, levonorgestrel IUS, etonogestrel implant).for one week following study drug administration.
3. Breastfeeding
4. Patients receiving concurrent ketamine therapy or who have received ketamine therapy during the trauma admission.
5. UDS screen on admission (if obtained) positive for alcohol, opioids other than prescribed for pain or maintenance opioids for OUD, or other substances of abuse
6. History of psychedelic substance use in the preceding 5 years
7. History (or active) cardiovascular disease (non-optimized coronary vascular disease, stable or unstable angina, new onset EKG abnormalities, congenital long QT syndrome, cardiac trauma involving surgical repair or CABG within 1 year)
8. Screening blood pressure SBP >140 mmHg or DBP > 90 mmHg on three separate occasions
9. Head trauma, traumatic brain injury, or concussion.
10. Tachycardia defined as HR > 100, averaged over the previous 12 hours, excluding intra-operative care)
11. History of dementia
12. History of pre-existing neurological conditions (including TIA, stroke, epilepsy, MS, ALS, Guillain-Barre, Parkinson's)
13. Patients on SSRIs, TCAs, MAO-Is, lithium, or other serotonergic medications, antipsychotics. Prohibited medications need to be discontinued at least 30 days prior to psilocybin dosing.
14. Patients that received intra-operative intravenous methadone dosing > 20 mg.
15. On vasopressors
16. Hepatic impairment, mild to moderate, with Child-Pugh score ≥ 7
17. Nicotine dependence, which would prevent the patient from staying in their room for the duration of the 8-hour psilocybin study period.
18. On sedating IV infusions (propofol, ketamine, fentanyl, benzodiazepine, dexmedetomidine)
19. History of suicidal or homicidal ideations within the last year
20. History of seizure disorder
21. Requiring restraints or active sitter
22. Patients with a history of poorly controlled anxiety (GAD7 score of 10 or more), poorly controlled depression (PHQ9 score of 15 or more), panic disorder, paranoia, PTSD, bipolar disorder, any primary psychotic disorder like schizophrenia, schizoaffective disorder, or antisocial personality disorder; personal or first- or second-degree relative history of psychotic or bipolar I or II disorder
23. History of Hallucinogen Use Disorder or Hallucinogen Persisting Perception Disorder (per DSM-V)
24. Unable to consent (intubated/sedated)
25. Intellectual disability
26. Additional or anticipated surgeries within 7248 hrs of psilocybin administration
27. Discharge from hospital pending within 24 hrs of psilocybin administration
28. Any allergy to psilocybin or other inert substances in the product

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Recruitment | From enrollment and receipt of psilocybin to 3 days post-treatment.
  Recruitment feasibility will be assessed by calculating the enrollment rate, defined as the number of participants enrolled and receiving psilocybin divided by the number of individuals determined eligible. Accrual rate will be calculated as total enrolled participants divided by the number of months recruitment occurred.
Feasibility: Retention | Day 5 post-treatment
  Retention will be calculated as the proportion of enrolled participants who receive treatment and complete required study assessments through follow-up day 5, divided by the number of individuals enrolled, treated, and not withdrawn. Feasibility target: ≥90% retention by day 5.
Feasibility: Completion of One-Month PROs | at 1-month post-treatment
  Feasibility will also be assessed by determining the completion rate of patient-reported outcome assessments 1 month after treatment, defined as the number of participants completing PROs divided by the number of enrolled participants who have not withdrawn. Feasibility target: ≥80% PRO completion at 1-month follow-up.

SECONDARY OUTCOMES:
Inpatient post-psilocybin acute pain scores (Visual Analogue Scale) | at baseline and Days 1, 2, 3, 5, and 7 after psilocybin administration
  Inpatient post-psilocybin acute pain scores assessed by visual analogue scale pain scores (VAS scores 0-10). Postoperative pain intensity assessed using a Visual Analogue Scale (VAS) ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst possible pain.
Opioid consumption | at baseline, and days 1, 2, 3, 5, and 7 after psilocybin administration.
  Opioid consumption measured in morphine milligram equivalents (MME), collected from the electronic medical record during hospitalization and after discharge.
Psilocybin Adverse side effects | measured at days 1, 2, 3, 5, 7 after psilocybin administration.
  Incidence and severity of adverse events following psilocybin administration, assessed through continuous clinical observation during the monitored dosing period, vital sign monitoring, and electronic medical record review.
Generalized Anxiety Disorder (GAD) | at Baseline, and 1-month after psilocybin administration
  Severity of anxiety symptoms assessed using the Generalized Anxiety Disorder-7 (GAD-7) scale. The GAD-7 consists of 7 items scored from 0 to 3, yielding a total score range of 0 to 21. Scores of 5, 10, and 15 represent mild, moderate, and severe anxiety, respectively. Higher scores indicate greater anxiety severity.
Physical Function (PROMIS Physical Function) | at Baseline and 1-month after psilocybin administration
  Physical function assessed using the PROMIS Physical Function instrument. Scores are reported as standardized T-scores with a mean of 50 and a standard deviation of 10. Higher scores indicate better physical function.
Resilience (Connor-Davidson Resilience Scale 10-Item Version) | Baseline and 1-month after psilocybin administration
  Resilience assessed using the 10-item Connor-Davidson Resilience Scale (CD-RISC-10). The CD-RISC-10 consists of 10 items evaluating an individual's ability to cope with stress and adversity. Each item is scored from 0 (not true at all) to 4 (true nearly all the time), yielding a total score range from 0 to 40. Higher total scores indicate greater resilience.
Depressive Symptoms (PHQ-9) | Baseline, and 1-month after psilocybin administration
  Patient-reported depressive symptom severity assessed using the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 consists of 9 items scored from 0 to 3, yielding a total score range of 0 to 27. Higher scores indicate greater severity of depressive symptoms.
PROMIS Pain Interference | Baseline, and 1-month after psilocybin administration
  Pain interference assessed using the PROMIS Pain Interference Short Form 8a. The instrument includes 8 items rated on a 5-point Likert scale from 1 (not at all) to 5 (very much). Raw scores are summed and converted to standardized T-scores with a mean of 50 and a standard deviation of 10. Higher T-scores indicate greater pain interference.
Post-psilocybin opioid-related harms | Measured at 1-month after psilocybin administration
  Occurrence of opioid-related harms following psilocybin administration, including unintended hospital admissions related to opioid use, opioid overdose events (fatal or non-fatal), opioid use disorder relapse, and emergency department visits related to opioid adverse events. Assessed by participant self-report and/or medical record review.

CONTACTS AND LOCATIONS:
Overall Officials: Trent D. Emerick, Principal Investigator — University of Pittsburgh / UPMC
Locations (1):
- UPMC Presbyterian, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No